CLINICAL TRIAL: NCT06852300
Title: Enhancing Concussion Assessment: A Multimodal Approach Using Neurocognitive Testing, Balance Evaluation, and Functional Near-infrared Spectroscopy
Brief Title: Sport-Related Concussion Recovery in Athletes
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Central Arkansas (Other)
Responsible Party: Principal Investigator, Hyung Rock Lee, Associate Professor, University of Central Arkansas
Other Study IDs: ERI19-141
Record Dates: First submitted 2025-02-11; First posted 2025-02-28 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-11

CONDITIONS: Concussion Mild; Concussion, Brain
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Concussed and Matched control Pool: The concussed group consists of collegiate athletes who have been diagnosed with a sport-related concussion by healthcare providers and meet the specified inclusion criteria. Injured participants will undergo testing within 72 hours of the injury and at predetermined time points post-concussion. Matched control participants will be assessed at the same time intervals as their injured counterparts to ensure comparability.
  The concussion test battery will comprise five assessments designed to evaluate sport-related concussion: 1. Health Questionnaire, 2. Sport Concussion Assessment Tool (SCAT), 3. Vestibular Ocular Motor Screening (VOMS) 4. Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT), 5. Balance Assessment.
  Additionally, the NIRSIT scanner will be utilized at each testing session to assess cognitive function and brain activity through Functional Near-Infrared Spectroscopy (fNIRS).
  Interventions: Device: Concussion Assessment Battery
- Pre-season and Post-Season Subject Pool: Participants will complete baseline concussion testing upon initiation into their intercollegiate athletic program. This group will consist of uninjured collegiate athletes from both contact and non-contact sports. Testing will be conducted at two time points: pre-season and post-season.
  Interventions: Device: Concussion Assessment Battery

INTERVENTIONS:
Device: Concussion Assessment Battery — The conclusion test battery will comprise five assessment designed to evaluate sport-related concussion:
  1. Health Questionnaire - Including as assessment of signs and symptoms.
  2. Sport Concussion Assessment Tool (SCAT)
  3. Vestibular Ocular Motor Screening (VOMS)
  4. Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT)
  5. Postural stability assessment (NeuroCom VSR Sport).
  Functional Neuroimaging Functional Near-Infrared Spectroscopy (fNIRS) is a non-invasive neuroimaging technology that measures brain activity by detecting changes in blood oxygenation. The NIRSIT scanner will be employed at each testing session to assess cognitive function using the Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) and postural stability using the NeuroCom VSR Sport system.

SUMMARY:
The goal of this study is to enhance the accuracy and sensitivity of concussion evaluation by integrating traditional assessment tools with emerging neuroimaging technologies, such as Functional Near-Infrared Spectroscopy (fNIRS). By systematically collecting data across multiple assessment domains-including sideline evaluations, neurocognitive testing, balance assessments, vestibular/ocular-motor screening (VOMS), and brain activity measurements-this study aims to improve the diagnostic process and ensure a safer return-to-play protocol for athletes recovering from sport-related concussions.

Research Questions:

1. How do traditional concussion assessment tools (SCAT, computerized neurocognitive tests, balance tests, and VOMS) compare to fNIRS in detecting changes in brain function following a sport-related concussion?
2. What is the relationship between pre-injury baseline measures, acute post- injury assessments, and recovery-phase evaluations in athletes diagnosed with a sport-related concussion?
3. Can fNIRS improve the sensitivity and specificity of concussion diagnosis compared to existing clinical assessments?
4. How do clinical symptoms, medical history, and other individual factors influence concussion recovery and return-to-play timelines?
5. Does integrating fNIRS with traditional assessment tools enhance the ability to track recovery progression and inform return-to-play decisions?

This study provides a comprehensive evaluation of concussion diagnosis and recovery while assessing the added value of fNIRS technology in improving clinical decision-making.

DETAILED DESCRIPTION:
1. Study Description This study aims to enhance the accuracy of concussion evaluation and improve return-to-play decisions for athletes recovering from sport-related concussions. By incorporating both traditional assessment tools and advanced neuroimaging technology, such as Functional Near-Infrared Spectroscopy (fNIRS), this research seeks to refine how concussions are diagnosed and monitored.
2. Who is Participating?

   College athletes will be recruited as part of their routine concussion baseline testing. Participants will include:
   * Athletes diagnosed with a sport-related concussion by healthcare providers.
   * Matched control athletes who have not sustained a concussion, assessed on the same schedule as concussed athletes.
   * Contact and non-contact sport athletes who have not experienced head injuries, tested before and after the season.
3. How is the Study Conducted?

   Testing occurs at four key time points:
   * Pre-Season (Baseline): Athletes complete a series of tests to establish their normal cognitive and physical function before any injuries occur.
   * Post-Injury (Within 72 Hours and Asymptomatic): If an athlete sustains a concussion, they undergo assessments shortly after the injury to measure its immediate effects.
   * Return-to-Play: Once the athlete has completed the necessary recovery steps and is cleared to return to play, they are reassessed to evaluate their recovery progress.
   * Re-Baseline (Six Months Post-Injury): Concussed athletes undergo follow- up testing at least six months after the injury to assess long-term recovery and determine whether any persistent neurophysiological changes remain.
4. What is Being Measured?

   This study utilizes a comprehensive concussion evaluation approach that includes:
   * Sideline assessments (e.g., Sports Concussion Assessment Tool [SCAT])
   * Computerized neurocognitive testing (Immediate Post-Concussion Assessment and Cognitive Testing)
   * Objective balance tests (NeuroCom VSR Sport)
   * Vestibular/Ocular-Motor Screening (VOMS)
   * Functional Near-Infrared Spectroscopy (fNIRS) to measure brain activity non-invasively
   * Clinical symptom tracking and medical history review
5. Why is This Study Important? The data collected will contribute to a robust database aimed at improving concussion assessment methods. By integrating fNIRS with standard concussion tests, this research seeks to enhance diagnostic accuracy, improve the ability to track recovery, and ensure a safer return to play for athletes. Additionally, the inclusion of a re-baseline assessment at six months post-injury will provide valuable insight into the long-term effects of concussion, informing future guidelines for concussion management. Ultimately, these findings could lead to more reliable tools for healthcare providers managing sport-related concussions.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited from athletes who have sustained a concussion and/or mild traumatic brain injury (mTBI), as determined by a physical examination conducted by medical staff based on the established concussion definition: biomechnical forces, typically resulting from a direct blow to the head, face, neck, or elsewhere on the body with an impulsive force transmitted to the head.

Exclusion Criteria:

* Current diagnosis of a psychiatric illness, attention deficit disorder, or learning disability.
* Current use of psychoactive medications.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited through university-affiliated sports medicine providers. When a student-athlete, including intramural sports participants, exhibits any signs, symptoms, or behaviors consistent with a sport-related concussion, they will be removed from practice or competition by either a member of the coaching staff or the sports medicine staff.
  Upon confirmation of a concussion diagnosis by the medical staff, the concussed athlete will be selected as a study participant and will be required to follow the post-concussion protocol outlined by the participating institution, which adheres to NCAA standards.
  Whenever possible, control subjects will be recruited from the same team, other sports teams, and/or students at the participating university who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-04-11 (Actual); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Prefrontal Cortex Activation during Neurocognitive Test using Functional Near- Infrared Spectroscopy (fNIRS) in Division-I Athletes following Sports-Related Concussion | From enrollment to 1 year after becoming asymptomatic.
  To compare prefrontal hemodynamic activation using fNIRS during the performance of a computerized ImPACT in a sample of concussed Division-I athletes tested within 72 hours post-injury compared to age-matched healthy subjects.
Prefrontal Cortex Activation During Postural Stability Testing Using Functional Near-Infrared Spectroscopy (fNIRS) in Division-I Athletes Following Sport-Related Concussion | From enrollment to 1 year after becoming asymptomatic
  The purpose of this study is to examine prefrontal cortex activation during postural stability testing in Division-I athletes following a sport-related concussion using functional near-infrared spectroscopy (fNIRS).
Evaluating the Sensitivity and Specificity of a Multifaceted Concussion Assessment Battery: A Comparison with Functional Near-Infrared Spectroscopy (fNIRS) Outcomes | From enrollment 1 year after becoming asymptomatic

SECONDARY OUTCOMES:
Enhancing Concussion Assessment Battery: Evaluating the Validity of Reliable Change Indices (RCI) in Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) using Machine Learning Approaches. | From enrollment 1 year after becoming asymptomatic
  Computerized neurocognitive tests like Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) are becoming more widely used by sports medicine professionals to evaluate concussions. A baseline ImPACT test is often recommended to help compare post-injury results, providing a more accurate picture of an athlete's cognitive function after a concussion. One method ImPACT uses to assess changes in cognitive function is the Reliable Change Index (RCI), which helps determine whether a difference in scores is meaningful. However, RCI has limitations, such as being less sensitive to real cognitive changes and the potential for misinterpretation. This study explores how machine learning approaches could improve the accuracy of concussion assessments using ImPACT scores.
Exploratory Structural Equation Modeling (ESEM) and Bifactor-ESEM analysis of the Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) symptom inventory. | From enrollment 1 year after becoming asymptomatic
  The Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) includes a symptom inventory widely used to assess self-reported concussion symptoms in athletes. This study will only use the self-reported symptom scale from the ImPACT as the primary Outcome Measure, with no other sub-scores or assessments included. The ImPACT symptom scale includes 22 symptoms rated on a 0 to 6 severity scale, with 0 indicating no symptom and 6 indicating the most severe. The total symptom score, ranging from 0 to 132, will serve as the primary Outcome Measure. Higher scores indicate greater symptom severity. This study will apply Exploratory Structural Equation Modeling (ESEM) and bifactor-ESEM to examine the factor structure, evaluate general and specific symptom dimensions, and improve the interpretability of ImPACT symptom scores for more accurate clinical assessments.
Neurocognitive Composite Scores and Symptom Scale Scores from the Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT): Traditional vs Remote Administration | From enrollment 1 year after becoming asymptomatic
  ImPACT is a widely utilized tool for assessing the cognitive function of collegiate athletes. Previous research has demonstrated that cognitive performance may vary depending on the environment in which concussion assessments are conducted.
  The ImPACT test battery consists of the following components administered in sequential order: (1) Demographics, (2) Symptom Scale, (3) Word Memory, (4) Design Memory, (5) X's and O's, (6) Symbol Match, (7) Color Match, (8) Three Letters, (9) Word Memory Delayed Recall, and (10) Design Memory Delayed Recall. All tests are automatically scored by the software.
  During the COVID-19 pandemic, many student-athletes transitioned from traditional, in-person concussion assessments to remote, at-home testing. This study aims to determine whether remote testing yields results comparable to traditional testing, ensuring the accuracy and consistency of concussion assessments regardless of the testing environment.

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Rock Lee, Ph.D, Principal Investigator — University of Central Arkansas
Locations (1):
- University of Central Arkansas, Conway, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided